CLINICAL TRIAL: NCT05120089
Title: Muscle Energy Technique Versus Myofacial Release in Adolescents With Spinal Deformity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant. Professor of physical therapy, Department of Physical Therapy for Pediatrics, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: muscle energy technique
Record Dates: First submitted 2021-09-17; First posted 2021-11-15 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Idiopathic Spinal Deformities
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- muscle energy technique (Experimental): Muscle energy technique is an associate degree of osteopathic manipulation methodology. The muscles of patients were used, on request, to type a singular controlled position, in a very specific direction, and against a distinctly executed therapist-applied counterforce. Muscle energy technique could be a post-isometric relaxation, because it reduces the tone of a muscle or cluster of muscle after a brief period following an isometric contraction. The result of post-isometric relaxation is mediated by receptive input from Golgi connective tissue organ (GTO) that has associate degree repressive result on the antagonist muscles mediated by the muscle spindle receptive. The technique will be applied for three month (3 session/week)
  Interventions: Other: muscle energy technique and myofacial release (physiotherapy techniques)
- myofacial release (Experimental): The technique will be applied for three month (3 session/week). All participants underwent ipsilateral side bending in a side-lying position, with the goals being de-rotation and scoliosis reduction.
  Interventions: Other: muscle energy technique and myofacial release (physiotherapy techniques)

INTERVENTIONS:
Other: muscle energy technique and myofacial release (physiotherapy techniques) — Each technique will be applied for three month (3 session/week)

SUMMARY:
Spinal deformity may not only alter the physical appearance, but may also have a psychological impact on the child, particularly in the adolescent to whom self- image is so important.

This study will investigate the effect of muscle energy technique compared to myofacial release in the adolescent with spinal deformities( scoliosis and/ or kyphosis).

ELIGIBILITY:
Inclusion Criteria:

* Children in this group will be healthy category according to CDC (Centers for Disease Control and Prevention) growth chart which ranged from BMI-for-age 5th to 85th percentiles . All children are normal &perform all activities of daily living
* They were able to understand and follow verbal commands and instructions included in the testing procedures.

Exclusion Criteria:

* All of them could be part of recreational activities in their public schools but no competitive sports. Children who participated in any regular sport activities involving the lower extremities will be excluded.
* None of them had any surgical intervention .
* None of them had any history of other musculoskeletal deformities or neuromuscular disorders.
* hey had neither visual, auditory defect.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
cobb angle for spinal deformities (scoliosis and/or kyphosis) | immediately before the beginning of the intervention procedures
  It is defined as the greatest angle at a particular region of the vertebral column, when measured from the superior endplate of a superior vertebra to the inferior endplate of an inferior vertebra. However, the endplates are generally parallel for each vertebra, so not all sources include usage of a superior versus inferior endplate in the definition.
cobb angle for spinal deformities (scoliosis and/or kyphosis) | by the end of successful three month of intervention
  It is defined as the greatest angle at a particular region of the vertebral column, when measured from the superior endplate of a superior vertebra to the inferior endplate of an inferior vertebra. However, the endplates are generally parallel for each vertebra, so not all sources include usage of a superior versus inferior endplate in the definition.

CONTACTS AND LOCATIONS:
Locations (1):
- AAA, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publishing by 12 month